CLINICAL TRIAL: NCT00542581
Title: Evaluation of the Acrysof Toric SN60T3 Intraocular Lens in Patients With Predicted Residual Corneal Astigmatism Between 0.75 and 1.00 D.
Brief Title: Acrysof Toric SN60T3corneal Astigmatism Between 0.75 and 1.00 D.
Acronym: TORILIOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SEI 07-001
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2010-10

CONDITIONS: Cataracts
Keywords: Visual Outcomes; Patient Satisfaction; Ophthalmology; Cataractous Lens
MeSH Terms: conditions — Cataract; Patient Satisfaction

ARMS (1):
- The Acrysof toric SN60T3 IOL (Experimental): Multifocal Intraocular Lens
  Interventions: Device: The Acrysof toric SN60T3 IOL

INTERVENTIONS:
Device: The Acrysof toric SN60T3 IOL — Intraocular Lens

SUMMARY:
The purpose of this study is to evaluate the visual outcomes and patient satisfaction after implantation of a toric IOL in patients with predicted residual corneal astigmatism between 0.75 and 1.00 D.

Cataract is prevalent throughout the world and IOLs are routinely implanted after the extraction of the cataractous lens. It is the most frequently performed surgery in the United States with an estimated 2-3 million procedures performed annually. With the aging population on the rise, as well as the increasing popularity of refractive intraocular lenses, the number of intraocular surgeries continues to rise. Over the years, the surgical technique has evolved from intracapsular extraction to modern phacoemulsification. This development has helped with the evolution of IOLs as well. The IOLs have advanced extensively: different materials and designs are available, permitting implantation through smaller, sutureless incisions. Traditional IOLs are of monofocal design providing vision at one distance, typically far; and correct mainly the spherical component of the refractive error. However, there are patients with corneal astigmatism that require additional surgical treatment such as laser correction (laser in situ leratomileusis, LASIK; photorefractive keratectomy, PRK) or limbal relaxing incisions, RLI). Another alternative is the use of a toric IOL, which has been especially designed to correct both the sphere and the astigmatism. The ACRYSOF Toric IOL is intended for primary implantation in the capsular bag of the eye for visual correction of aphakia and preexisting comeal astigmatism in adult patients with or without presbyopia, who desire improved uncorrected distance vision, reduction of residual refractive cylinder and increased spectacle independence for distance vision.

The treatment selection of the corneal astigmatism depends on the amount of cylinder as follows, between 0.25 and 0.75 D creating the surgical incision on the steep axis; between 0.75 and 1.75 D, RLI; between 1 and 2.25 D, toric IOLs; and between 1 and 3.00 D, LASIK/PRK.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, unmasked pilot study.

1. SETTING: Storm Eye Institute, Medical University of South Carolina, Charleston, SC and one additional site in USA.
2. SUBJECTS A total of 40 eyes (20 per site) of 20 subjects of both sexes and any race undergoing routine phacoemulsification and intraocular lens implantation will be included.

   2.1. Patient Inclusion Criteria: Subjects MUST fulfill the following conditions to qualify for enrollment into the trial 2.1.1. Subject must have an age-related cataract in both eyes.

   2.1.2. 21 years of age or older. 2.1.3. Patient must desire cataract extraction. 2.1.4. Expected maximum of 2 weeks and minimum of 1-week interval between first and second eye surgeries. 2.1.5. Cross-cylinder value calculation from the Toric Calculator indicates a cross-cylinder correction from 0.75D to 1.0D in at least one eye and up to 1.75 in the fellow eye.

   2.1.6. Willing and able to comply with scheduled visits and other study procedures.

   2.2. Patient Exclusion Criteria: Subjects with ANY of the following conditions on the eligibility exam may NOT be enrolled into the trial.

   2.2.1. Preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmus or macrophthalmus, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc. 2.2.2. Planned postoperative refraction for mono-vision. 2.2.3. Uncontrolled diabetes. 2.2.4. Use of any systemic or topical drug known to interfere with visual performance.

   2.2.5. Contact lens use during the active treatment portion of the trial. 2.2.6. Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.

   2.2.7. Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control. 2.2.8. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results. 2.2.9. Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial. 2.2.10. Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye. 2.2.11. Other ocular surgery at the time of the cataract extraction.

   The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates the patient is unsuitable for the trial.

   2.3. Surgical Exclusion Criteria

   The study lens should not be implanted and the patient should be excluded from the study if any of the following complications are encountered during surgery:

   2.3.1. Significant anterior chamber bleeding. 2.3.2. Detached Descemet's membrane 2.3.3. Iris damage 2.3.4. Inability to achieve secure, symmetric, "in the bag" position of the IOL: posterior capsule rupture, radial tear in capsulorhexis, vitreous loss, zonular rupture.

   2.3.5. Use of corneal sutures for more than 1 week.

   2.4. Post-implantation Exclusion Criteria 2.4.1. Haptic not in the capsular bag. 2.4.2. Decentration of the IOL of more than 1.0 mm 2.4.3. Ocular pathologies potentially affecting visual acuity that were not evident prior to surgery.

   The principal investigator reserves the right to declare a patient ineligible or nonevaluable based on medical evidence that indicates the patient is unsuitable for the trial.
3. STUDY ENROLLMENT PROCEDURES Subjects will be recruited from the corneal and anterior segment clinic at Storm Eye Institute and satellite offices. Once identified as a study candidate, the patient will be asked if he/she would like to participate. A study coordinator or one of the investigators will answer any and all questions and will obtain informed consent. The patient will understand that participation in the study will not affect their quality of care.
4. STUDY INTERVENTION The Acrysof toric SN60T3 IOL is approved by the Food and Drug Administration (FDA).

   The examinations and treatments used in this protocol are similar to those used in routine practice. Therefore, the additional risks involved in this study are extremely low. Patients will undergo routine cataract extraction and intraocular implantation of the Acrysof toric lens in both eyes.
5. STUDY VISIT SCHEDULE AND ASSESSMENTS (Table 1) 5.1. Visit Schedule

Patients will be examined at the following intervals:

1. Visit 1: Preoperative evaluation completed not more than four weeks before surgery
2. Visit 2: Date of Surgery
3. Visit 3: 14 ± 2 days postoperative
4. Visit 4: 30 ±5 days postoperative
5. Visit 5: 90 ±7 days postoperative
6. Visit 6: 180 ±10 days postoperative Additional office visits as required for medical safety. On such visits an unscheduled patient visit case report should be completed.

6. MEASUREMENTS AND EVALUATIONS

6.1. Visit 1: Preoperative assessment included a thorough medical history and a complete eye examination. The latter will include ETDRS uncorrected distance visual acuity (UCDVA), manifest refraction, ETDRS best corrected distance visual acuity (BCDVA), slit-lamp exam, manual keratometry, Orbscan, and a quality of vision questionnaire will be evaluated as well. Informed consent is to be obtained prior to performing the procedures in this study. Patient must review and sign the documentation. Women of childbearing potential will undergo a pregnancy test and will only be entered into the trial if this is negative.

6.2. Visit 2: Surgery will be performed by the surgeon under topical anesthesia. A standard phacoemulsification and posterior chamber lens insertion will be performed according to the investigator's preferred technique. If a major complication occurs during surgery (e.g. expulsive hemorrhage or vitreous loss requiring vitrectomy), the patient will be excluded from the trial. Subjects will be implanted with the Acrysof Toric SN60T3 IOL. Postoperatively, patients will be instructed to follow the standard of care routinely used after cataract extraction.

6.3. Visits 3, 4 and 5: On postoperative days 30 ±5, 90 ±7 and 180 ±10, ophthalmic examination to include: UCDVA, BCDVA, manifest refraction, slit lamp biomicroscopy, IOL position from slit lamp evaluation, manual keratometry and Orbscan. Absolute residual cylinder will be evaluated as well as change in axis orientation (determined by the postoperative manifest refraction), and distance spectacle independence.

Table 1. Study Assessments

Visit 1 Preop Visit 2 Date of surgery Visit 3 Day 30 ±5 Visit 4 Day 90 ± 7 Visit 5 Day 180 ± 10 Inclusion & exclusion criteria X Signed informed consent X Demographics X Symptoms Assessment X X X X UCVA X X X X Manifest Refraction X X X X BCVA X X X X Manual keratometry X X X X Orbscan X X X X Intraocular pressure X Slit lamp examination X X X X Dilated fundus exam X Quality of vision and distance vision spectacle independence questionnaire X X X X Adverse events X X X X X

7. STATISTICAL CONSIDERATIONS

7.1. Sample size calculation: This is a pilot study.

7.2. Statistical Method: All data will be collected by the study coordinators. Data will be entered into an Access database. The database will be password protected and access will be restricted to study personnel. Data analysis will be performed without patient identification. Comparisons and statistical analysis will be done to determine if any statistical differences exist between preoperative and postoperative visits. Statistical analysis will be done using standard descriptive statistics and other tests as deemed appropriate based on the distribution of the data. If data is normally distributed, test such as the t-test will be used, while non-normally distributed data will be analyzed using the Wilcoxon test for comparison between the groups. ANOVA and Kruskal-Wallis tests will be used for comparison between baseline and postoperative visits. A P less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST fulfill the following conditions to qualify for enrollment into the trial

* Subject must have an age-related cataract in both eyes.
* 21 years of age or older.
* Patient must desire cataract extraction.
* Expected maximum of 2 weeks and minimum of 1-week interval between first and second eye surgeries.
* Cross-cylinder value calculation from the Toric Calculator indicates a cross-cylinder correction from 0.75D to 1.0D in at least one eye and up to 1.75 in the fellow eye.
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

Subjects with ANY of the following conditions on the eligibility exam may NOT be enrolled into the trial.

* Preoperative ocular pathology:

  * Amblyopia
  * Rubella cataract
  * Proliferative diabetic retinopathy
  * Shallow anterior chamber
  * Macular edema
  * Retinal detachment
  * Aniridia or iris atrophy
  * Uveitis
  * History of iritis
  * Iris neovascularization
  * Medically uncontrolled glaucoma
  * Microphthalmus or macrophthalmus
  * Optic nerve atrophy
  * Macular degeneration (with anticipated best postoperative visual acuity less than 20/30)
  * Advanced glaucomatous damage, etc.
* Planned postoperative refraction for mono-vision.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* Pregnant or nursing mothers and females of childbearing potential not practicing a reliable and medically acceptable method of birth control.
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye.
* Other ocular surgery at the time of the cataract extraction.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary benefit from implantation of an IOL and participation in this study is the restoration of useful vision following removal of the cataracts. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D. Solomon, MD, Principal Investigator — Storm Eye Institute
Locations (1):
- Medical Unvirsity of South Carolina, Charleston, South Carolina, United States